CLINICAL TRIAL: NCT00383500
Title: To Prospectively Evaluate the Potential for Simple, Effective Lymphedema Prophylaxis in Breast Cancer Survivors Who Show Early Evidence of High-risk Status
Brief Title: Lymphedema Prophylaxis in Breast Cancer Survivors Who Show Early Evidence of High-risk Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley Rockson, Professor of Lymphatic Research and Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-01671; 95970 (Other: Stanford University Alternate IRB Approval Number); BRSNSTU0007 (Other: OnCore Number)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Lymphedema; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Flexitouch device (Experimental): Participants will self-administer lymphedema management via daily use of the Flexitouch device, an intermittent pneumatic compression device (aka, lymphedema pump)
  Interventions: Device: Flexitouch
- Manual Lymphatic Drainage (MLD) (Experimental): Participants will self-administer lymphedema management via daily manual lymphatic massage therapy, using a Class 1 compression garment
  Interventions: Device: Class 1 compression garment
- Observational Control (no intervention) (No Intervention): Control group, no intervention. No Flexitouch or manual massage therapy

INTERVENTIONS:
Device: Flexitouch — A standard of care intermittent pneumatic compression device (aka, lymphedema pump)
  Other Names: Tactile Systems Technology, Inc.; Biocompression; Lymphatic massage therapy
  Arms: Flexitouch device
Device: Class 1 compression garment — Manual lymphatic drainage therapy to provide lymphatic massage, using a Class 1 compression garment supporting the arm during heavy exercise or where the risk of trauma maybe increased (ie, flight, elevation, etc).
  Other Names: Manual lymphatic drainage; Lymphatic massage therapy
  Arms: Manual Lymphatic Drainage (MLD)

SUMMARY:
To compare the effectiveness of usual treatments for lymphedema [massage and elastic compression sleeve, instituted at-risk and before the development of swelling (lymphedema)], compared to the use of a newly-marketed device, the Flexitouch, which electronically simulates the effect of massage upon lymph flow.

DETAILED DESCRIPTION:
The current investigation is designed to prospectively evaluate the potential for simple, effective lymphedema prophylaxis in breast cancer survivors who show early evidence of high-risk status. There is growing evidence that the mechanisms of lymphatic repair after injury are mediated through lymphatic flow. Accordingly, this study assess if physical measures designed to prophylactically augment lymphatic flow after surgical interventions for breast cancer (eg, Flexitouch and manual lymphatic massage) will reduce the incidence of lymphatic stagnation, assessed as incidence of lymphedema, when compared to patients who receive conventional "watch and wait" interventions (observation).

The specific aims of the study are

1. to prospectively assess the presence of newly developing lymphedema in each study subgroup through serial assessment of segmental interstitial fluid content by multiple frequency bioimpedance
2. to evaluate the preventive interventions in a prospective, randomized fashion, contrasting the responses of equivalent numbers of patients randomized to 2 experimental arms and the control arm of the study
3. to correlate the bioimpedance findings with concurrently derived, serial assessments of limb volume

Recent advances in the medical understanding of the biological processes of lymphatic development and repair suggest that these mechanisms may be able to be manipulated to enhance the regenerative responses in the lymphatic vasculature following injury. Breast cancer-associated lymphedema is a model of such an acquired form of lymphatic vasculature insufficiency. Clinically, this poses a substantial clinical problem. It is estimated at 1woman in 4 who survives a breast cancer intervention will develop lymphedema, often progressively. The appearance of lymphedema has documented adverse effects on physical and psychologically well-being. New insights into lymphatic repair suggest that such mechanisms can be employed in a prophylactic fashion to forestall or eliminate the development of lymphedema. This proposal investigates this hypothesis in a prospective fashion, using a randomized trial design in 80 patients enrolled at the time of breast cancer surgery. If the investigation documents a beneficial effect of preventive measures, it could have a profound impact on subsequent breast cancer care. These measures are simple and cost-effective and, could help to eliminate the impact of a substantial detractor to the improved longevity and health that breast cancer survivors otherwise may expect to enjoy.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral breast cancer
* Scheduled to undergo breast surgery and axillary lymph node dissection, with or without breast conserving techniques.
* Referred to the surgeons of the Stanford University Breast Cancer Program
* Capacity to provide informed consent.
* All experimental protocols will be reviewed and approved by the Stanford Institutional Review Board for the Protection of Human Subjects.

Exclusion Criteria:

* Other serious systemic illness (renal failure, hepatic dysfunction, congestive heart failure, neurological or psychological impairment) that would confound the study or impair the patients' ability to participate.
* Recurrent breast cancer or other forms of pre-existing lymphedema.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley G Rockson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced in May 2005 and concluded 13 March 2012. Subjects were recruited from the medical clinics and Stanford University Hospital and Clinics.
Groups:
- Flexitouch Device: Lymphedema management via Flexitouch device, an intermittent pneumatic compression device (aka, lymphedema pump)
- Manual Lymphatic Drainage (MLD): Lymphedema management via self-administered manual lymphatic massage therapy
- No Intervention Control: No intervention observational control
Period: Overall Study
Arm/Group | Flexitouch Device | Manual Lymphatic Drainage (MLD) | No Intervention Control
Started | 27 | 24 | 24
Completed | 19 | 21 | 22
Not Completed | 8 | 3 | 2
Not completed — Withdrawal by Subject | 8 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group I: This group of patients will receive the device.
- Group II: This group of patients will receive prophylactic MLD
- Group III: This is the control group; they will receive no treatment
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Total
Number analyzed (Participants) | 27 | 24 | 24 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 19 | 65
  >=65 years | 3 | 2 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 24 | 75
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 26 | 22 | 24 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 2 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 2 | 0 | 0 | 2
  White | 17 | 20 | 20 | 57
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Assessment of Lymphedema by Multiple Frequency Bioimpedance Spectroscopy
Description: Successful, serial multiple frequency bioimpedance assessment for newly developing lymphedema in the 3 study groups
Time Frame: 36 months
Population: All enrolled patients in the trial who did not withdraw or were lost to follow-up
Measure: Number; unit: participants
Groups:
- Manual Lymphatic Drainage (MLD): Lymphedema management via self-administered manual lymphatic drainage therapy
Arm/Group | Flexitouch Device | Manual Lymphatic Drainage (MLD) | No Intervention Control
Number analyzed (Participants) | 19 | 21 | 22
participants | 19 | 21 | 22

2. Primary Outcome: Incidence of Lymphedema (Newly-developing)
Description: Incidence of newly-developing lymphedema for each study cohort, as detected by serial multiple frequency bioimpedance spectroscopy scans for increased interstitial fluid within regional tissues.
Time Frame: 3 years of semi-annual follow-up
Measure: Number; unit: participants
Arm/Group | Flexitouch Device | Manual Lymphatic Drainage (MLD) | No Intervention Control
Number analyzed (Participants) | 19 | 21 | 22
participants | 1 | 5 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Flexitouch Device | Manual Lymphatic Drainage (MLD) | Observational Control (no Intervention)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 1/19 | 5/21 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexitouch Device (N=19) | Manual Lymphatic Drainage (MLD) (N=21) | Observational Control (no Intervention) (N=22)
Lymphedema (Vascular disorders) | 1 (1) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No